CLINICAL TRIAL: NCT07102030
Title: Subgrouping SLE - a New Approach to Understand the Pathogenesis and Improve Treatment
Acronym: SLEsubgroups
Status: Recruiting | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other); National Institutes of Health (NIH) (NIH); The Swedish Research Council (Other Government); Reumatikerförbundet (Unknown)
Responsible Party: Sponsor
Other Study IDs: VR 2022-00783
Record Dates: First submitted 2025-07-28; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Blood samples (serum, plasma, PAx tubes). DNA will be extracted. Urine and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- SLE patients: Patients fulfilling ACR 1982 or SLICC 2012 criteria for SLE. No interventions
- Controls: General population controls matched from the National Patient Registries for age, gender and area of living

SUMMARY:
The goal of this observational study is to investigate different phenotypes among patients with SLE and to compare with matched general population controls. The main questions we aim to answer are:

A To investigate if subgroups of patients with systemic lupus erythematosus (SLE) defined by autoantibodies, genetic predisposition or biomarkers, rather than the present diagnostic entities account for the high risk of premature vascular disease.

B To perform in depth studies of selected patient groups to shed light on the autoimmune mechanisms behind antiphospholipid (aPL) antibodies and nephritis and their association to vascular disease in SLE and APS Participants will be investigated in person by a nurse and a rheumatologist. Data on previous and present disease characteristics, anthropometric measurements and health related quality of life (according to selfreported questionnaires) will be entered into a data base. Blood samples (plasma serum and DNA), urine and saliva is stored in a corresponding biobank.

Researchers will compare identified subgroups of SLE patients to each other and to matched population controls.

DETAILED DESCRIPTION:
The clinical base for this application is a series of cross-sectional studies, performed every 10 years, including all consenting SLE patients at Rheumatology Karolinska. The first studies were initiated 1995-99, with second follow-up 2004-14. Since 2015, a third follow-up of prevalent and new cases is ongoing (presently comprising 400 patients, inclusions have been temporarily slowed by the Covid-19 pandemic). Very detailed clinical characterization, lifestyle questionnaires, together with results from carotid ultrasound and bone mineral density measures have been tabulated. General disease activity as well as features of lupus nephritis, and detailed autoantibody profiles are recorded at inclusion. Samples (plasma, serum, DNA, urine and saliva) are stored. We have a common database for the three cross-sectional studies. The total number of well-characterized SLE patients in these studies is today 867 SLE patients and >250 APS patients.

Population based controls identified in the national population registry (NPR), individually matched for age, sex, and residency have been investigated in person according to the same structured protocol (n=320). New controls will be included to match the "2015+ study".

ELIGIBILITY:
Inclusion Criteria:

SLE according to criteria (ACR82 or SLICC 2012) and consenting to participate

Exclusion Criteria:

Not possible to read and understand patient information due to language barriers or psychological/psychiatric disorders Not consenting

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SLE patients as described above who are cared for at karolinska University Hospital, Danderyds Hospital or Center forRheumathology (CFR) in Stockholm and matched general population controls
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2015-02-15 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Autoantibody defined subgroups | 2024- 2027
  Subgroups will be defined based on presence of autoantibodies
Cardiovascular events | 2024-2027
  Cardiovascular events will be collected during follow up in National Patient Registries

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Clinical and autoantibody data collected at inclusion
Supporting Information: Study Protocol, ICF, CSR
Time Frame: July 15 2025 until July 15 2027
Access Criteria: Selected data will be shared with Christian Lood, University of Washington USA, using Managed File Transfer at Karolinska Institutet.